CLINICAL TRIAL: NCT07327814
Title: Mental Calculus Can Enhance Gait Performance in Post-Stroke Patients: A Randomized Controlled Trial
Brief Title: Effect of Mental Arithmetic Priming on Gait and Balance in Stroke
Acronym: MA-Stroke
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lebanese University (Other)
Responsible Party: Principal Investigator, Ahmad Rifai Sarraj, Professor, Lebanese University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ED-STROKE-MENTAL-CALCULUS
Record Dates: First submitted 2025-12-25; First posted 2026-01-08 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Stroke; Hemiparesis; Gait Disorders; Posture; Disorders
Keywords: Stroke; Hemiparesis; Posture; Balance; Gait Disorders
MeSH Terms: conditions — Stroke; Paresis; Mobility Limitation; Disease

STUDY DESIGN:
Who Masked: Participant
Masking Description: Single Blind (Participant)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention: Behavioral: Mental Arithmetic (Experimental): Visual presentation of arithmetic equations (Addition, Subtraction, Multiplication) projected on a screen. Participants must calculate and verbally report the answer within a 10-second window per equation.
  Interventions: Behavioral: Mental Arithmetic
- Passive Viewing (Placebo Comparator): Passive viewing of a black screen with no cognitive demand.
  Interventions: Behavioral: Passive Viewing

INTERVENTIONS:
Behavioral: Mental Arithmetic — Visual presentation of arithmetic equations (Addition, Subtraction, Multiplication) projected on a screen. Participants must calculate and verbally report the answer within a 10-second window per equation.
  Arms: Intervention: Behavioral: Mental Arithmetic
Behavioral: Passive Viewing — Passive viewing of a black screen with no cognitive demand.
  Arms: Passive Viewing

SUMMARY:
This study investigates the effect of cognitive priming through mental arithmetic on functional mobility in post-stroke patients. It hypothesizes that performing mental calculations (addition, subtraction, multiplication) prior to movement stimulates frontoparietal networks, thereby improving gait speed and dynamic balance compared to a passive control condition.

DETAILED DESCRIPTION:
Stroke often results in impaired sensorimotor integration and executive dysfunction, leading to gait and balance deficits. Emerging evidence suggests a link between numerical cognition and motor control networks. This randomized controlled trial compares an experimental group (performing 30-second mental arithmetic tasks) against a control group (passive visual exposure). Functional mobility is assessed immediately following the cognitive stimulus using the Ten-Meter Walk Test (10mWT) and the Timed Up and Go (TUG) test to evaluate the immediate "priming" effects of cognitive load on motor performance.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of stroke.
* Mini-Mental State Examination (MMSE) score ≥ 23.
* Ability to walk 10 meters independently (with or without assistive device).

Exclusion Criteria:

* Hemianopia.
* Wernicke's aphasia or Global aphasia.
* Orthopedic injuries or recent surgeries affecting the lower limbs.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Estimated)
Dates: Start 2026-02-11 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Gait Speed (10mWT) | Immediately following the 30-second cognitive stimulus.
  Assessed using the Ten-Meter Walk Test (10mWT). Participants walk 14 meters; time is recorded for the middle 10 meters to determine steady-state gait speed.
Dynamic Balance (TUG) | Immediately following the 30-second cognitive stimulus.
  Assessed using the Timed Up and Go (TUG) test. Time taken to stand from a chair, walk 3 meters, turn, walk back, and sit down.

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) that underlie the results reported in this article (after de-identification) will be shared. This includes the data used to generate the tables and figures.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available beginning 6 months and ending 5 years following article publication.
Access Criteria: Data will be shared with researchers who provide a methodologically sound proposal to the corresponding author. Proposals should be directed to ahmadrifaisarraj@ul.edu.lb. To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Background] Khayat J, Champely S, Diab A, Rifai Sarraj A, Fargier P. Effect of mental calculus on the performance of complex movements. Hum Mov Sci. 2019 Aug;66:347-354. doi: 10.1016/j.humov.2019.05.008. Epub 2019 May 28. No abstract available. PMID 31146193